CLINICAL TRIAL: NCT05823441
Title: Effects of Oxytocin Nasal Inhalation and Social Familiarity on Empathy Analgesia: a Factorial Randomized Controlled Trial
Brief Title: Effect of Oxytocin Nasal Inhalation on Empathy Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Head of anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022PHD012-001
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Oxytocin; Pain; Empathy; Social Familiarity; Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OS group (Placebo Comparator): Half an hour after the volunteers inhaled 24 units of oxytocin spray, they watched the pre recorded video (attached with pictures and introductions of strangers) and underwent a pain test.
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Stranger
- PS group (Placebo Comparator): Half an hour after the volunteers inhaled the same amount of saline spray, they watched the pre recorded video (with pictures and introductions of strangers attached) and received a pain test.
  Interventions: Drug: Placebo; Behavioral: Stranger
- OA group (Experimental): Half an hour after the volunteers inhaled 24 units of oxytocin spray, they watched the pre recorded video (attached with pictures and introductions of acquaintances) and underwent a pain test.
  Interventions: Drug: Oxytocin nasal spray; Behavioral: Acquaintance
- PA group (Placebo Comparator): Half an hour after the volunteers received the same dose of saline, they watched the pre recorded video (attached with pictures and introductions of acquaintances) and received the pain test.
  Interventions: Drug: Placebo; Behavioral: Acquaintance

INTERVENTIONS:
Drug: Oxytocin nasal spray — Volunteers inhale 24 units of oxytocin spray
  Arms: OA group; OS group
Drug: Placebo — Volunteers inhale 24 units of placebo spray
  Arms: PA group; PS group
Behavioral: Stranger — Volunteers watch a video of a pain test and attach a photo of a stranger
  Arms: OS group; PS group
Behavioral: Acquaintance — Volunteers watch a video of a pain test and attach a photo of an acquaintance
  Arms: OA group; PA group

SUMMARY:
This study recruited healthy volunteers and randomly divided them into four groups. They inhaled oxytocin or saline, and watched a pain test video with photos of acquaintances or strangers, respectively, to test whether their feelings of the same thermal pain stimulus had changed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* During pregnancy;
* Have participated in any research related to pain;
* Sleep disorders;
* Used alcohol, caffeine, nicotine, or other psychoactive substances within 24 hours before the test;
* Experienced intense pain requiring medical analgesia within three months prior to the trial;
* Taking any medication, including over the counter medication;
* Addiction to alcohol, tobacco, or drugs;
* A history of any respiratory, circulatory, neurological, musculoskeletal, and/or mental illness;
* Current symptoms of depression and/or anxiety. (See quantitative sensor testing for specific standards)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
NRS score | Half an hour after inhaling spray
  numerical rating scale of pain， ranging from 0 = "no pain" to 10 = "the most intense pain that is tolerable".

SECONDARY OUTCOMES:
EEG | about 3 hours
  Frequency of electroencephalogram
Brief Profile Of Mood States | about 3 hours
  Brief Profile Of Mood States is a 30 item self-report psychological instrument intended for use with adults age 18 and above. Response format consisted of the following 5-point Likert scales: 0：not at all; 1：a little; 2：moderately; 3：quite a bit; and 4：extremely.
Beck Depression Inventory | about 3 hours
  Beck Depression Inventory
WLEIS-C | about 3 hours
  The English version of the scale was developed by Wong and Law and used as an evaluation tool for emotional intelligence level surveys, the Chinese version of emotional intelligence level consists of 16 items scale (WLEIS-C) , including self-emotional perception (4 items), others' emotional perception (4 items), emotional control (4 items), emotional use (4 items) 4 Dimensions, a total of 16 items. Using Likert 7-level scoring method, '0' stands for 'very disagree' and '6' stands for 'very agree'. The higher the score, the higher the emotional intelligence level.
STAI | about 3 hours
  state-trait anxiety inventory
BES-C | about 3 hours
  Chinese version of Basic Empathy Scale.The scale was divided into two dimensions: emotional empathy, which comprised 11 items, and cognitive empathy, which comprised nine items, yielding a total of 20 items (including eight reverse-scoring items). A five-point Likert scale was used, where 1 = "completely disagree" and 5 = "completely agree." A high score indicated strong empathy.
The Positive and Negative Affect Scale | about 3 hours
  is a 20 item self-report psychological instrument，contains 10 items for positive and 10 items for negative emotions. All the items are rated on a scale ranging from 1 ("very slightly or not at all") to 5 ("extremely").
NRS score | about 3 hours
  numerical rating scale of pain， ranging from 0 = "no pain" to 10 = "the most intense pain that is tolerable".

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China